CLINICAL TRIAL: NCT02264197
Title: Single-dose Pharmacokinetics of 160 mg BIBX 245 CL and Effect of Food After Oral Administration of Tablets to Healthy Subjects (Randomized, 2-way-cross-over, Open Study)
Brief Title: Investigation of Pharmacokinetics of BIBX 245 CL and Safety in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 537.7
Record Dates: First submitted 2014-10-14; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- BIBX 245 CL - fed (Experimental): after a light breakfast with 40 g fat
  Interventions: Drug: BIBX 245 CL - fed
- BIBX 245 CL - fasted (Active Comparator)
  Interventions: Drug: BIBX 245 CL- fasted

INTERVENTIONS:
Drug: BIBX 245 CL - fed
  Arms: BIBX 245 CL - fed
Drug: BIBX 245 CL- fasted
  Arms: BIBX 245 CL - fasted

SUMMARY:
Aim of this trial is to investigate the single dose pharmacokinetics and the effect of food on single dose of 160 mg 245 CL (two 80 mg tablets) as well as its safety

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 50 years
* Broca >= -20% and <= +20%

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurologic disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (<= 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (<= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation > 100 ml (<= 4 weeks prior to administration or during the trial)
* Excessive physical activities (<= 10 days prior to administration or during the trial)
* Any laboratory value outside the reference range or clinical relevance

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 1998-05; Primary Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum measured concentration of the analyte in plasma) | up to 24 hours post dose
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours post dose
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 24 hours post dose
λz (Terminal rate constant in plasma) | up to 24 hours post dose
t½ (Terminal half-life of the analyte in plasma) | up to 24 hours post dose
MRTtot (Mean residence time) | up to 24 hours post dose

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 20 days
Assessment of tolerability by investigator | after 20 days